CLINICAL TRIAL: NCT02849730
Title: Postoperative Pain and Patient-controlled Epidural Analgesia Related Adverse Effects in Young and Elderly Patients
Brief Title: Epidural PCA Related Adverse Effects in Young and Elderly
Status: Completed | Type: Observational
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Dr. Koh, Jae Chul, MD, Assistant professor, Department of Anesthesiology and Pain medicine, Severance Hospital
Other Study IDs: 2016-0295-001
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Pain, Postoperative
Keywords: Epi-PCA; Patient controlled analgesia; Epidural patient controlled analgesia; Elderly patient; Side effect; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Young adults: Patients aged 20 to 39 who had used fentanyl/ropivacaine based Epi-PCA for postoperative pain.
  Interventions: Device: Fentanyl/ropivacaine based Epi-PCA
- Elderly patients: Patients aged 70 and over who had used fentanyl/ropivacaine based Epi-PCA for postoperative pain.
  Interventions: Device: Fentanyl/ropivacaine based Epi-PCA

INTERVENTIONS:
Device: Fentanyl/ropivacaine based Epi-PCA — Fentanyl and ropivacaine was diluted and administered to the patients according to the clinician's determination. The clinician decided dose, infusion rate, bolus dose, lockout time and total amount of drug mixed in the Epi-PCA.
  Other Names: Epidural patient controlled analgesic device

SUMMARY:
In this retrospective study, postoperative pain score, epidural patient controlled analgesia (Epi-PCA) related complications, the risk factors for requirement of rescue analgesics and antiemetics will be evaluated in young and elderly patients, respectively, using fentanyl and ropivacaine-based Epi-PCA during postoperative 48 hours after various surgeries.

DETAILED DESCRIPTION:
Since 2010, A PCA service team in the investigators' hospital have collected multidisciplinary clinical data from all the patients who used epidural-patient controlled analgesia (Epi-PCA) postoperatively in aim of the assessment of clinical outcome. The investigators reviewed the collected data from the patients who had used Epi-PCA for pain control after an elective surgery under general or spinal anesthesia between Sep. 2010 and Nov. 2015. The need for informed consent was waived for this study. For the Epi-PCA, fentanyl and ropivacaine was diluted and administered to the patients according to the clinician's determination.

The data of the PCA regimen which has been decided were recorded and analyzed. Demographic variables including age, sex, body mass index, American Society of Anesthesiologists (ASA) physical status and history of smoking, motion sickness, postoperative nausea/vomiting, hypertension and diabetes mellitus will be analyzed. Anesthesia and surgery-related variables including the duration of anesthesia, the type of anesthesia (general or spinal), laparoscopy and the operation site (categorized in abdominal, thoracic, upper & lower extremities, head & neck, spine and others) will be also analyzed. PCA-related variables including total dose of fentanyl for two days (µg/kg), use of mixed additional analgesics and antiemetics in PCA and discontinuation of PCA will be analyzed. Postoperative variables including the numeric rating scale (NRS, 0-10, 0 = no symptom; 10= unthinkable worst pain) for pain, requirements of rescue analgesics and antiemetics will be analyzed. In addition, the postoperative complications including nausea, vomiting, headache, dizziness, and sedation will be analyzed. All the recorded postoperative variables at post-anesthesia care unit, 6-12, 12-18, 18-24 and 24-48 hrs after anesthesia will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had used Epi-PCA for pain control after an elective surgery under general or spinal anesthesia between Sep. 2010 and Nov. 2015.

Exclusion Criteria:

* Age < 20 years old,
* Age 40 to 69,
* Routine use of analgesics/antiemetics
* Imperfect data

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Collected data from the patients who had used Epi-PCA for pain control after an elective surgery under general or spinal anesthesia between Sep. 2010 and Nov. 2015.
Sampling Method: Non-Probability Sample
Enrollment: 2435 (Actual)
Dates: Start 2016-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Rescue Analgesics Requirement | Postoperative up to 48 hours
  The percentage of patients who required rescue analgesics at least once during the postoperative 48-hour period
Incidence of discontinuation of Epi-PCA | Postoperative up to 48 hours
  The percentage of patients who discontinued Epi-PCA

SECONDARY OUTCOMES:
Postoperative Pain in Numeric Pain Scale | Postoperative up to 48 hours
  The Numeric Pain Scale (NRS - 0: no pain, 10: worst pain can't imagine) for pain measured once at each time periods (0~6, 6~12, 12~18, 18~24, 24~48 hours)
Incidence of Nausea and Vomiting | Postoperative 48 hours
  The percentage of participants who had nausea and vomiting during postoperative 48 hours
Incidence of Dizziness or Headaches | Postoperative up to 48 hours
  The percentage of participants who had headache and dizziness during postoperative 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dong Woo Han, MD, PhD, Study Chair — Gang Nam Severance Hospitial
Locations (1):
- Gangnam Severance hospital, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No